CLINICAL TRIAL: NCT03814850
Title: Remote Ischemic PreConditioning Provides Neuroprotection: A Phase 2, Single Center, Randomized, Double-Blind, Sham-Controlled, Safety and Efficacy Study Evaluating the Use of Remote Ischemic Preconditioning in Patients Undergoing Endovascular Repair of Brain Aneurysms
Brief Title: Remote Ischemic PreConditioning (RIPC)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were identified per inclusion/exclusion criteria
Sponsor: Sebastian Koch (Other)
Responsible Party: Sponsor-Investigator, Sebastian Koch, Professor of Clinical Neurology, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20191282; 20180869 (Other: University of Miami IRB)
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Unruptured Cerebral Aneurysm
Keywords: brain aneurysm; endovascular repair; ischemic stroke
MeSH Terms: conditions — Intracranial Aneurysm; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person performing the RIPC is not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group: standard blood pressure cuff (Experimental): A standard blood pressure cuff inflated on the participants arm for 4 cycles; each cycle will include 5 minutes of inflation followed by 5 minutes of deflection. RIPC will be applied via a standard blood pressure cuff. The ischemic cycle will involve cuff inflating to 30mmHg above resting systolic blood pressure and demonstration of loss of radial pulse.
  Interventions: Device: Standard Manual Aneroid Sphygmomanometer
- Sham group: standard blood pressure cuff (Sham Comparator): The blood pressure cuff will be inflated to 30mmHg during the first 5 minutes of each cycle and deflated for the following 5 minutes, with re-demonstration of radial pulse. This will be repeated for 4 cycles.
  Interventions: Device: Standard Manual Aneroid Sphygmomanometer

INTERVENTIONS:
Device: Standard Manual Aneroid Sphygmomanometer — Use of a standard manual blood pressure cuff and manometer for the conditioning intervention.

SUMMARY:
The purpose of this study is to learn about protecting the brain from low blood flow (ischemia) with limb preconditioning. From human studies the investigators know that the brain can be protected from dangerous low blood flow by reducing the blood flow to an arm or leg for just a short period of time. This is called limb preconditioning. The investigators are studying the safety and feasibility of preconditioning and their effect of protecting the brain from ischemia in two different groups. This is a Phase 2, randomized, double-blind, sham-controlled, design. Up to 50 male and female patients undergoing elective endovascular repair of unruptured brain aneurysm who are randomized to the remote ischemic preconditioned or sham group will be enrolled. This study consists of one 3-9 month study period for each patient plus up to 14 days for enrollment activities. Subjects are required to return between 3-9 months for end-of-study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of an unruptured brain aneurysm deemed suitable for repair by neuroendovascular techniques involving intraluminal occlusion by detachable platinum coils, stent-assisted coiling, pipeline stent, balloon-assisted coiling, covered stent only, neck-bridge device, re-coiling, or re-treatment of a previously coiled/treated aneurysm. There are no restrictions on adjunctive devices.
2. Absence of ongoing ischemic symptoms such as transient ischemic attacks, minor strokes, stroke-in-evolution, or clinical evidence of cerebral vasospasm within 2 weeks prior to randomization. (If a CT scan, cerebral angiogram, or other imaging performed during the 2 weeks prior to randomization shows radiological vasospasm deemed by the treating physician to be potentially clinically significant, the subject is excluded).
3. Male or female with a minimum age of 18 years on the day of enrollment.
4. Informed consent and availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.

Exclusion Criteria:

1. Dissecting or mycotic brain aneurysm. Fusiform or atherosclerotic intracerebral aneurysms may be eligible for the trial if endovascular treatment is planned with a goal of exclusion of the aneurysm from the circulation.
2. Planned endovascular vessel sacrifice as the primary modality for aneurysm treatment.
3. Known history of life-threatening allergic reaction to any medication.
4. Soft tissue, orthopedic, or vascular injury which, in the judgment of the investigator, would preclude arm ischemic conditioning (e.g. superficial wounds, venous, arterial ulcers, gangrene).
5. History of peripheral vascular disease or deep vein thrombosis in either arm.
6. Women who are pregnant, or have a positive urine or blood (β-hCG) pregnancy test.
7. Women who are breastfeeding.
8. Any clinically significant psychiatric or psychological disease, which would preclude the patient from completing the protocol.
9. Pre-morbid (estimated) modified Rankin scale score of greater than 2. A subject is not excluded if they have a pre-morbid modified Rankin scale of greater than 2 but the disability does not interfere with the subject's ability to complete an MRI and the cognitive evaluations.
10. Previous serious traumatic brain injury that would preclude the patient from completing the protocol or preclude MRI analysis of small strokes.
11. Patients with peripherally inserted central catheters, hemodialysis shunts, arteriovenous fistulae or grafts in the treatment limb, or lymphedema.
12. Patients with known Human Immunodeficiency Virus (HIV) infection.
13. Patients who are unable to have an MRI scan for any reason.
14. Participation in a clinical trial with an investigational drug within 30 days preceding this study. Previous participation in any clinical trial investigating ischemia following endovascular aneurysm treatment, participation in another trial involving RIPC, or prior receipt of RIPC.
15. Severe or unstable concomitant condition disease or chronic condition, which, in the opinion of the investigator, could affect assessment of the safety or efficacy of study intervention.
16. Any other medical condition that the site investigator deems would put the patient at excessive risk of participation in the study or an expected life expectancy less than 1 year or that would result in inability to collect clinical outcomes at 30 days.
17. Systolic blood pressure above 200mm Hg.
18. Cannot tolerate inflation of the tourniquet on their arm consistent with blood pressure cuff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all adverse events and serious adverse events. | 9 months
  Adverse events are all conditions/symptoms/findings and all abnormal clinically significant laboratory tests both expected and unexpected, occurring from onset of the intervention until study completion.
Change in procedurally-induced vascular cognitive impairment. | Baseline, Day 2-4
  As measured by the NIH-toolbox for neurocognitive testing.NIH-Toolbox normalized scores to define a single cognitive battery index.C. Score:0= No deficit, no change; 400= Maximum deficit.

SECONDARY OUTCOMES:
Change in procedurally-induced vascular cognitive impairment. | Baseline, 3-9 months.
  As measured by the NIH-toolbox for neurocognitive testing. NIH-Toolbox normalized scores to define a single cognitive battery index.C. Score:0= No deficit, no change; 400= Maximum deficit
Volume of embolic strokes by Diffusion Weighted Imaging (DWI). | Timeframe: Baseline, 12-96 hours post procedures
  Measured in select patients by Diffusion Weighted Imaging (DWI) via Magnetic Resonance Imaging (MRI) that undergo 4 cycles of 5 minutes of limb ischemia followed by 5 minutes reperfusion.
Volume of embolic strokes by Fluid-attenuated Inversion Recovery (FLAIR). | Timeframe: Baseline, 12-96 hours post procedures.
  Measured in select patients by Fluid-attenuated Inversion Recovery (FLAIR) via Magnetic Resonance Imaging (MRI) that undergo 4 cycles of 5 minutes of limb ischemia followed by 5 minutes reperfusion.
Frequency of large (>10 cc value) strokes. | 2-4 days post procedures.
  As measured by MRI imaging when performed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Starke, M.D., Principal Investigator — University of Miami; Sebastian Koch, MD, Study Director — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No